CLINICAL TRIAL: NCT03832699
Title: Oral Dydrogesterone vs. Vaginal Micronized Progesterone for Luteal Phase Support in Frozen-thawed Embryo Transfer: a Non-inferiority Randomized Clinical Trial
Brief Title: Oral Dydrogesterone vs. Vaginal Micronized Progesterone for Luteal Phase Support in Frozen-thawed Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, Principal investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0013-19-WOMC
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: ART
MeSH Terms: interventions — Dydrogesterone; Progesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral progesterone (Experimental)
  Interventions: Drug: Dydrogesterone 10 MG
- Vaginal progesterone (Active Comparator)
  Interventions: Drug: Endometrin 100Mg Vaginal Insert

INTERVENTIONS:
Drug: Dydrogesterone 10 MG — Oral progesterone 10 mg TID
  Arms: Oral progesterone
Drug: Endometrin 100Mg Vaginal Insert — Vaginal Endometrin 100 mg twice daily
  Arms: Vaginal progesterone

SUMMARY:
The current trial is intended to assess the efficacy of oral versus vaginal progesterone for luteal support in frozen IVF cycles.

DETAILED DESCRIPTION:
Progesteron is used for luteal phase support in IVF cycles. Progesterone can be administered vaginally and orally. Duphaston is an oral progesterone drug, which has recentlly been proven effective in fresh cycle IVF. Yet, less is known regarding its efficacy in frozen cycle IVF. Thus, the objective of our trial is to compare the efficacy of vaginal and oral progesterone in frozen IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-39
* Modified natural cycle (induction of ovulation with HCG)
* Consent to participation

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Up to 9 months
  Birth of a live infant after 24 weeks gestation

SECONDARY OUTCOMES:
Clinical pregnancy rate | Outcome assesed 6-7 weeks following treatment
  Viable pregnancy as demonstrated by ultrasound
Implantation rate | Outcome assessed 6-7 weeks following treatment
  Number of gestational sacs divided by number of embryos transferred (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Ganer Herman, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel